CLINICAL TRIAL: NCT04301947
Title: Acute Effect of a Gluteal Activation Warm-up on Hip Muscle Activity and Kinematics During a Single Leg Squat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Caroline Ruschel, Professor Ruschel, Caroline, University of the State of Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE24886619400000118
Record Dates: First submitted 2020-02-05; First posted 2020-03-10 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hip Adduction; Gluteus EMG Activity
Keywords: single leg squat; 2D kinematics; hip adduction; EMG; gluteal activation; warm-up

STUDY DESIGN:
Intervention Model Description: This is a descriptive quantitative study with cross-over design of repeated measures.The study will be conducted in two stages. In the first stage, anthropometric data collection, intervention protocol application and biomechanical data collection will be performed. The intervention application order will be random and counterbalanced which half of the participants will receive the gluteal pre-activation protocol and the other half a standard warm-up protocol at the first visit. In the second stage, the intervention will be applied and biomechanical data will be collected. In this context, the following routine will be performed: (1) Preparation and familiarization (2) intervention protocol application (standard warm-up or gluteal pre-activation) (3) Immediately after the protocol, three (3) repetitions of the single-legged squat will be performed and (4) data collection of maximal voluntary isometric contraction will be extracted.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All participants enrolled will receive instructions about the protocols by the same investigator. An independent researcher will perform block randomization, with a 1:1 allocation ratio and allocation order (using the random list generator at www.randomization.com). The results will be stored in sequentially numbered opaque sealed envelopes that will be opened before the first intervention in the presence of the participant. An independent investigator will code the data and make it available to the investigator who applied the intervention after a wash-out period for processing. The processed data will be sent to this independent researcher, who will decode it and perform the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard warm-up protocol (Active Comparator): The standard warm-up protocol consists of 5 (five) minutes of stationary cycling, followed by calf, hamstring and quadriceps stretching. For all stretching positions 30 (thirty) seconds will be set. For calf stretching, the participant places his hands on the waist and projects his dominant limb behind of the center of mass line, the contralateral limb will be placed forward until the stretch sensation on the dominant limb start. For hamstring stretching, the participant will be instructed to bend over the hip, reaching the foot of the dominant limb in dorsiflexion. Emphasis will be placed on maintaining the heel of the dominant limb on the floor and maintaining posture. Finally, for quadriceps stretching, the participant will perform a knee flexion and will hold the dominant lower limb foot close to the gluteus with the ipsilateral upper limb hand. Emphasis will be placed on maintaining trunk posture.
  Interventions: Other: Standard warm-up protocol
- Gluteal activation warm-up (Experimental): The gluteal activation warm-up protocol consists of performing a standard warm-up protocol with additional "shell" exercise. The shell exercise will be performed with the participant side-lying with hip and knee flexed, an elastic band (PREFORM BETTER Inc. Rhode Island, USA) will be placed around the distal thigh to promote resistance and the participants will be instructed to perform hip abduction movements. The exercise will be performed in multiple sets (3 sets) of 12 repetitions, with 30 seconds interval between exercises in order to minimize the fatigue effect. Medium and heavy elastic bands tensions will be used and adjusted according to the effort perception parameter from the OMNI scale for effort perception for resistance training.
  Interventions: Other: Gluteal activation warm-up protocol

INTERVENTIONS:
Other: Standard warm-up protocol — Stationary cycling and lower limb stretching exercises
  Arms: Standard warm-up protocol
Other: Gluteal activation warm-up protocol — Standard warm-up protocol + Clam exercise (3 sets of 12 repetitions each)
  Arms: Gluteal activation warm-up

SUMMARY:
Gluteal activation warm-up is one of the modalities being investigated recently. Although widely used in clinical and sports practice, it is unclear whether, in fact, performing gluteal activation exercises in warm-up is effective in increasing electromyographic activation (EMG), as well as the mechanisms that explain eventual gluteal activation improvement of neuromuscular function. Thus, the aim of this study is to verify the acute effect of a gluteal activation warm-up protocol on gluteus maximus (superior fibers) and gluteus medius EMG activation and kinematics during single leg squat. The hypotheses of this study are that after a gluteal activation warm-up program, there will be an increase in the muscle recruitment (mean) levels of the gluteus maximus (superior fibers) and gluteus medium. About kinematics, the hypotheses is that a decrease on hip adduction absolute angle and hip and knee frontal plane ROM on maximum knee flexion during single leg squat will occur. Physically active adults from 18 to 35 years old, with no history of previous injury or surgery on the lower limbs, who present excessive hip adduction during single-leg squat on the dominant limb in previous evaluation via visual scoring scale will participate in this study. The design adopted will be performed in the following order: (1) Preparation and familiarization. (2) Intervention protocol (standard warm-up protocol or the gluteal activation warm-up protocol), (4) immediately after the intervention protocol, the subjects will perform 3 single-leg squats and (5) EMG and MIVC strength test. The standard warm-up consist 5 minutes on a stationary bike and 30 seconds calf, hamstrings and quadriceps stretch. The gluteal activation warm-up protocol consists of performing the standard warm-up protocol and 3 sets of 12 repetitions clam exercise, using a elastic band (Perform Better®, USA). Exertion perception will be controlled using an exertion perception scale (OMNI). From kinematic and EMG data, absolute values of the hip adduction, hip and knee ROM in the frontal plane of the dominant limb and mean EMG activation data from the gluteus maximus (superior fibers) and gluteus medius muscles we will extracted, respectively. All data will be analyzed using descriptive and inferential statistics. (p <0.05).

DETAILED DESCRIPTION:
Muscle pre-activation is the application of exercises to specific muscle groups performed in the warm-up phase in order to increase the neuromuscular response. Among different modalities of warm-up, gluteal activation warm-up is one of the modalities being investigated recently. The hip joint perform movements in the three planes of movement (sagittal, frontal and transverse), being the gluteus maximus and gluteus medius the main muscles that perform triple actions in this joint. Not only about the joint itself but, the research about the hip joint kinematics is of interest due to its importance on pelvic stability and trunk control, playing a key role on motor control during dynamic tasks. This also claim for the increase emphasis that has been put on strategies that could help clinicians to better understand factors associated with hip muscle dysfunction and injury occurrence. The literature has been shown that hip muscle weakness are associated with the occurrence of knee injuries like ACL (anterior cruciate ligament) tears or patellofemoral dysfunction and interventions focused on better activate hip muscles, specifically gluteus maximus and medium, have been demonstrating to be key strategies to reduce undesirable movement patterns associated to lower limb injury risk factors. Although widely used in clinical and sports practice, it is unclear whether, in fact, performing gluteal activation exercises in warm-up phase is effective in increasing electromyographic activation (EMG), as well as the mechanisms that explain eventual gluteal activation improvement of neuromuscular function. Thus, the aim of this study is to verify the acute effect of a gluteal activation warm-up protocol on gluteus maximus (superior fibers) and gluteus medius EMG activation and kinematics during single leg squat. The hypotheses of this study are that after gluteal activation warm-up program, there will be an increase in the muscle recruitment (mean) levels of the gluteus maximus (superior fibers) and gluteus medium. About kinematics, the hypotheses that a decrease on hip adduction absolute angle and hip and knee frontal plane ROM (range of motion) on maximum knee flexion during single leg squat will occur. Participants will perform the test procedures during two visits, with a minimum interval of 24 hours and maximum of one week. The study will be conducted in two stages. In the first stage, anthropometric data collection, intervention protocol application and biomechanical data collection will be performed. The intervention application order will be random and counterbalanced which half of the participants will receive the gluteal gluteal activation warm-up protocol and the other half a standard warm-up protocol at the first visit. In the second stage, the intervention will be applied and biomechanical data will be collected. In this context, the following design will be adopted on both days: (1) Preparation and familiarization (2) intervention protocol application (standard warm-up or gluteal activation warm-up) (3) Immediately after the protocol, three (3) repetitions of the single leg squats will be performed and (4) data collection of maximal voluntary isometric contraction will be extracted. Since the first visit, the participant's routine will be performed as follow: (1) Anamnesis; (2) Anthropometric assessment; (3) electromyography electrodes fixation; (4) retro-reflective markers fixation for kinematic evaluation. (5) intervention protocol execution; (6) Assessment of movement pattern during single leg squats and (7) evaluation of muscle strength by handheld dynamometry and muscle electrical activity by electromyography via maximal voluntary isometric contraction (MIVC). The participants will be invited to make a second visit to the laboratory, to be scheduled in advance, to repeat the procedures for assessing muscle strength, muscle electrical activity, performing another intervention protocol and assessing kinematic during the single leg squat. At first, participants will receive all information about the procedures. For all tests, participants will receive specific positioning and execution guidance. For the anamnesis, participants will answer general questions about past and current health history, dominant lower limb and physical exercise through a questionnaire. For anthropometric data, measurements of height and body mass will be performed. For EMG and kinematic, electromyography electrodes will be fixed to the region of the gluteus maximus and gluteus medius muscles in the hip for assessment of electrical activity and retro-reflexive markers will be placed on anatomical marks of interest (lower limbs and pelvis) to evaluate the kinematic on single leg squat. A intervention protocol will be decided by draw and familiarization will be given informing position and execution of the exercises. Immediately after the intervention protocol, a single leg squat test will be performed only on the dominant limb. For such, three consecutive trials will be performed, without intervals between them. Familiarization and information will be given about the performance of the test. Kinematic data will be processed using KINOVEA software (Creative Commons 3.0, France). From the reference points attached only on the dominant limb, four body segments will be virtually reconstructed: pelvis, thigh, leg and foot. From these segments, the angles will be calculated at a static position, representing the start position and deepest knee flexion degree representing the end of the movement. The absolute values of hip adduction at maximum knee flexion angle (primary outcome) and differences between the two moments (ROM) in each test will be calculated to obtain the following ranges of motion (secondary outcome): knee on sagittal plane (flexion / extension), knee on frontal plane (adduction / abduction), hip on frontal plane (adduction / abduction) and pelvis on frontal plane (pelvic drop / contralateral elevation). All the three squat repetitions will be analyzed. The average of the three repetitions will be used for statistical analysis. EMG raw signals will be assessed using an TeleMyo DTS Desk Receiver® electromyograph (Noraxon® USA, Inc., Scottsdale, AZ, USA). Data will be sent in real time to a computer via Bluetooth, recorded and analyzed by MyoResearch 3.6 Applications Clinical software (Noraxon USA, Inc., Scottsdale, AZ, USA). A 10-500 Hz bandpass filter will be applied to EMG data. The MIVC with maximum amplitude of the EMG signal during the MIVC of each muscle will be recorded and will represent 100% of muscle activity. Muscle activities recorded during squats will then be expressed as a percentage of MVIC.

For statistical analysis, a IBM SPSS Statistics software, version 20.0 (IBM Corporation, Armonk, New York) will be utilized to process and calculate data. A descriptive analysis of anthropometric variables will be performed to characterize the subjects, mean and standard deviation will be adopted for numerical variables. For inferential statistics, tests for normality will be employed. From kinematic data, only absolute values of hip frontal angle and ROM for hip and knee on frontal plane (hip and knee adduction/abduction) and knee on sagittal plane (knee flexion/extension) will be calculated. For EMG, mean EMG activity (Gluteus maximus and medius) over the three single leg squat repetitions will be considered for statistical analysis. Data reliability between conditions will be based on the intraclass correlation coefficient (ICC).

ELIGIBILITY:
1. Inclusion criteria:

   * Age: between 18 and 35 years old.
   * Physically active: regularly participating in activities of training sessions 3x/week and minimum 20 minutes duration for each session.
   * No complaints about pain or musculoskeletal impairment on dominant leg during the first contact/interview.
   * Pelvic drop presentation during single leg squat on dominant leg: Will be included only those participants who, on the first interview, present excessive hip adduction during the single-leg squat task detected by visual assessment screening.
2. Exclusion criteria:

   * History of recent upper limb or spine injury.
   * Surgery on dominant limb or time less than one year of surgery on non dominant limb.
   * Complaints about cardiovascular or systemic diseases that could limit performance of the tests.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pre standard warm-up protocol hip adduction | two minutes before the intervention
  Absolute angle of hip adduction at peak knee flexion during squat leg squat, expressed in degrees (º).
Post standard warm-up protocol hip adduction | two minutes after the intervention
  Absolute angle of hip adduction at peak knee flexion during squat leg squat, expressed in degrees (º).
Pre gluteal activation warm-up protocol hip adduction | two minutes before the intervention
  Absolute angle of hip adduction at peak knee flexion during squat leg squat, expressed in degrees (º).
Post gluteal activation warm-up protocol hip adduction | two minutes after the intervention
  Absolute angle of hip adduction at peak knee flexion during squat leg squat, expressed in degrees (º).

SECONDARY OUTCOMES:
Pre standard warm-up protocol gluteus maximus and medius EMG activity. | two minutes before the intervention
  Mean neuromuscular activity at moments of interest (maximum knee flexion) for each muscle (gluteus maximus and gluteus medium), expressed as a percentage of MIVC (%MIVC)
Post standard warm-up protocol gluteus maximus and medius EMG activity | two minutes after the intervention
  Mean neuromuscular activity at moments of interest (maximum knee flexion) for each muscle (gluteus maximus and gluteus medium), expressed as a percentage of MIVC (%MIVC)
Pre gluteal activation warm-up protocol gluteus maximus and medius EMG activity. | two minutes before the intervention
  Mean neuromuscular activity at moments of interest (maximum knee flexion) for each muscle (gluteus maximus and gluteus medium), expressed as a percentage of MIVC (%MIVC)
Post gluteal activation warm-up protocol gluteus maximus and medius EMG activity. | two minutes after the intervention
  Mean neuromuscular activity at moments of interest (maximum knee flexion) for each muscle (gluteus maximus and gluteus medium), expressed as a percentage of MIVC (%MIVC)

OTHER OUTCOMES:
Pre standard warm-up protocol hip and knee adduction/abduction and knee flexion range of motion | two minutes before the intervention
  Difference of the angles of hip and knee on the frontal plane and knee on the sagittal plane between static position and peak knee flexion, expressed in degrees (º).
Post standard warm-up protocol hip and knee adduction/abduction and knee flexion range of motion | two minutes after the intervention
  Difference of the angles of hip and knee on the frontal plane and knee on the sagittal plane between static position and peak knee flexion, expressed in degrees (º).
Pre gluteal activation warm-up protocol hip and knee adduction/abduction and knee flexion range of motion | two minutes before the intervention
  Difference of the angles of hip and knee on the frontal plane and knee on the sagittal plane between static position and peak knee flexion, expressed in degrees (º).
Post gluteal activation warm-up protocol hip and knee adduction/abduction and knee flexion range of motion | two minutes after the intervention
  Difference of the angles of hip and knee on the frontal plane and knee on the sagittal plane between static position and peak knee flexion, expressed in degrees (º).

CONTACTS AND LOCATIONS:
Overall Officials: CAROLINE RUSCHEL, PE PhD, Study Chair — University of the State of Santa Catarina; MARCELO P CASTRO, PT PhD, Study Director — Neuromusculoskeletal Rehab. and Clinical Biomechanics Laboratory - LaBClin
Locations (1):
- University of the State of Santa Catarina (UDESC), Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
authors declare that deidentified IPD that underlie the results in the publication, Study Protocol and Statistical Analysis Plan will be shared immediately following publication and ending three years after publication with investigators that intend to use data for research purposes, as approved by an independent review committee. Requests should be addressed to caroline.ruschel@udesc.br accompanied by the approved proposal.
Supporting Information: SAP
Time Frame: Immediately following publication and ending three years after publication.
Access Criteria: Investigators whose intention is to use the data for research purposes as approved by an independent review committee should direct the approved proposal to caroline.ruschel@udesc.br to request access.